CLINICAL TRIAL: NCT05070741
Title: Heat Shock Therapy to Improve Mitochondrial Function in Neuropathy
Acronym: HOTFUN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with study recruitment in target population. Subjects who were enrolled completed study activities.
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Paige Geiger, PhD, Professor of Molecular & Integrative Physiology, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00143811
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: PreDiabetes; Neuropathy
MeSH Terms: conditions — Prediabetic State | interventions — Diathermy

STUDY DESIGN:
Intervention Model Description: This prospective, observational cohort pilot study will recruit 20 patients with prediabetes with or without peripheral neuropathy (painful and non-painful) to participate in a 4-week heat therapy intervention. After screening, informed consent, and enrollment into the study, subjects will undergo a pre-intervention evaluation that will assess metabolic biomarkers and heat shock protein levels (blood), peripheral neuropathy, and epidermal evaluation (skin biopsy). After the skin biopsy has the appropriate time to heal (approximately 7-14 days), the subjects will undergo 45-minute heat treatments in 40°C water, three times weekly, for 4 weeks. After completion of heat treatments, subjects will undergo a repeated post-intervention evaluation and skin biopsy. Statistical approaches will compare pre- and post-heat therapy measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heat Therapy Treatment (Experimental): This study will recruit subjects to participate in heat therapy treatment at the University of Kansas Medical Center (KUMC). After pre-screening, informed consent, and enrollment, all subjects will have baseline laboratory assessments as well as an examination for neuropathy and a lower distal leg biopsy (3mm). Subjects will complete 12 heat therapy treatments over the course of 4 weeks. Within 24-48 hours after the last heat therapy experience, post-treatment laboratory assessments as well as an examination for neuropathy and a lower distal leg biopsy (3mm) will be performed.
  Interventions: Behavioral: Heat Therapy

INTERVENTIONS:
Behavioral: Heat Therapy — Subjects will undergo 12 hot water immersions of 40.5 degrees Celsius for approximately 45 minutes per session over 4 weeks. Subjects will be immersed up to the shoulder in a 40°C hot tub until rectal temperature (Tre) increases by 1°C (~20 minutes). Subjects will then remain in the water bath submerged to waist level to maintain Tre between 38.5 and 39.0°C for another 30 minutes (approx. total time submerged ~50 minutes). Following hot water immersion, subjects will be monitored for another 10 min, or until Tre falls below 38.5°C. Core temperature will be monitored using either 1) a rectal probe with sterile disposable sheaths or 2) a sterile disposable rectal thermistor probe (401 A/C, Advanced Industrial Systems, Inc., Harrods Creek, KY) to be inserted ~1 inch past the anal sphincter (inserted by participant). Heart rate and blood pressure will be monitored throughout the treatment. Subjects will be continually monitored and removed from the hot bath if Tre exceeds 39.5°C.

SUMMARY:
Sensory dysfunction as a result of peripheral nerve damage is a significant problem that leads to reduced quality of life for patients. The prevalence of sensory dysfunction in peripheral neuropathy associates with epidemic increases in prediabetes and diabetes, but also is relevant to chemotherapy treatments and genetic disorders. Clinical approaches to treat peripheral neuropathy and to stimulate axon growth in settings of peripheral axon loss are limited. Although new drugs will hopefully be forthcoming, the most promising approaches likely involve behavioral and lifestyle interventions. Mitochondrial dysfunction is emerging as a key cellular contribution to peripheral axon health and peripheral neuropathy. Mitochondrial deficiencies contribute to neuropathy and include impaired mitochondrial problems with trafficking, mitophagy, fission, and biogenesis. All of these are thought to lead to a bioenergetic crisis, ending in distal axonal degeneration, sensory dysfunction and pain. Heat shock proteins play a critically important role in cellular homeostasis and increasing heat shock protein functions within cells leads to a range of positive improvements, particularly in mitochondria. In addition, new evidence suggests that increasing heat shock protein responses in peripheral nerves has powerful, positive impacts on sensory function and neuropathy.

Our interdisciplinary team will investigate the role of mitochondrial dysfunction in peripheral neuropathy and translate these approaches to improve treatment for patients with peripheral neuropathy. The investigators hypothesize that novel heat treatment interventions that improve mitochondrial function will improve metabolic symptoms and peripheral nerve mitochondria, leading to improvements in sensory function, via heat shock protein induction. The investigators will employ immersion heat treatment to elevate heat shock protein responses that induce positive changes in peripheral nerve mitochondria. One aspect is to confirm the efficacy, safety, and potential for heat treatment to improve sensory dysfunction in human patients with prediabetes. The goal of this proposal is 1) to test the breadth of heat treatment on various forms of neuropathy, 2) identify mechanisms in which heat treatment improves mitochondrial function, and 3) test the efficacy, safety, and potential for heat treatment to improve sensory dysfunction in human patients with prediabetes.

ELIGIBILITY:
Inclusion criteria:

1. both males and females,
2. ages 45-75,
3. have suspected or diagnosed prediabetes with or without neuropathy (to be confirmed at pre-intervention evaluation).

Exclusion criteria:

1. skin conditions, circulatory insufficiency, or open wounds in the leg that would interfere with healing from a biopsy;
2. stroke or other significant nervous system pathology;
3. lidocaine allergy;
4. anticipated difficulty with blood clotting due to disorder or use of a blood thinner such as Coumadin, Xarelto, or Eliquis;
5. use of any medication used to treat abnormal blood glucose such as Metformin;
6. body weight > 350 lbs.;
7. history of anemia or vitamin b12 deficiency;
8. clinical anemia (hematocrit <32 for women, <36 for men);
9. abnormal SPEP result;
10. history of cancer or chemotherapy treatment;
11. current or recent use (within the last 6 months) of artificial fingernails / nail enhancements that would interfere with quantitative sensory testing;
12. no special classes of subjects such as fetuses, neonates, pregnant women, prisoners, institutionalized individuals, non-English speaking individuals, or other who may be considered vulnerable populations will be included in this study.

Withdrawal/Termination criteria: Prediabetes will be determined using the American Diabetes Association (ADA) Diabetes Management Guidelines. The subject will meet the criteria for a diagnosis of pre-diabetes if the subject has one or more positive test(s) for either A1c (5.7-6.4%), fasting glucose (100-125 mg/dl), or 2-hr oral glucose tolerance test (140-199 mg/dl). If at pre-intervention evaluation, the subject does not meet the criteria for prediabetes (lower than the above-mentioned range), meets the ADA criteria for diabetes (higher than the above-mentioned range), the subject will be considered a screen fail and will not progress to skin biopsy or intervention.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paige Geiger, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited for this study through flyers posted at the University of Kansas Medical Center, in the community, and electronically via websites and email. Participants were also recruited utilizing the Frontiers Research Participant Registry. Participants were offered a $25 for completing Visits 1, 2, 15 and 16; and $15 for completing Visits 3-14; after completing each of the visits ($280 total) to aid with time and transportation.
Groups:
- Heat Therapy Treatment: Subjects will undergo 12 hot water immersions of 40.5 degrees Celsius for approximately 45 minutes per session over 4 weeks. Subjects will be immersed up to the shoulder in a 40°C hot tub until rectal temperature (Tre) increases by 1°C (~20 minutes). Subjects will then remain in the water bath submerged to waist level to maintain Tre between 38.5 and 39.0°C for another 30 minutes (approx. total time submerged ~50 minutes). Following hot water immersion, subjects will be monitored for another 10 min, or until Tre falls below 38.5°C. Core temperature will be monitored using either 1) a rectal probe with sterile disposable sheaths or 2) a sterile disposable rectal thermistor probe (401 A/C, Advanced Industrial Systems, Inc., Harrods Creek, KY) to be inserted ~1 inch past the anal sphincter (inserted by participant). Heart rate and blood pressure will be monitored throughout the treatment. Subjects will be continually monitored and removed from the hot bath if Tre exceeds 39.5°C.
Period: Overall Study
Arm/Group | Heat Therapy Treatment
Started | 3
Completed | 2
Not Completed | 1
Not completed — Failed initial laboratory testing and was unable to progress to heat therapy treatment. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 66 [65 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2
Pre-Diabetes [Count of Participants; unit: Participants] | 2
Neuropathy [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Fasting Blood Glucose (FBG)
Description: The study team will measure fasting blood glucose at baseline and post-intervention.
Time Frame: At baseline and post-intervention (~4-5 weeks after first visit)
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 2
mg/dL | -1 [-6 to 4]

2. Primary Outcome: Change in 2-hr Glucose
Description: The study team will measure 2-hr Glucose at baseline and post-intervention. To complete the oral glucose tolerance test (OGTT), the participant will drink a sweet, concentrated solution of glucose (Azer Scientific Glucola, 75 g) within 5 minutes. Afterwards, the participant will wait 2-hrs and blood will be drawn to test glucose and insulin levels.
Time Frame: At baseline and post-intervention (~4-5 weeks after first visit)
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 2
mg/dL | 23.5 [-24 to 71]

3. Primary Outcome: Change in Intraepidermal Nerve Fibers (IENF)
Description: The study team will count intraepidermal nerve fibers at baseline and post-intervention.
Time Frame: At baseline and post-intervention (~4-5 weeks after first visit)
Population: Study was terminated early due to difficulties with study recruitment in target population. Samples collected were not analyzed, and will never be analyzed, thus no data were collected for this Outcome Measure
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Quantitative Sensory Testing (QST) Scores
Description: Pressure pain sensitivity is measured by the Multimodal Automated Sensory Testing (MAST) System (measured at the thumbnail). It yields a pressure pain threshold value measured in kg/cm2.
Time Frame: At baseline and post-intervention (~4-5 weeks after first visit)
Measure: Number; unit: kg/cm2
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 2
kg/cm2 | -0.01

5. Secondary Outcome: Change in Concentration of Heat Shock Protein 72
Description: Serum levels of heat shock proteins (HSP72) will be measured via Western blots and Elisa assays in serum at baseline and post-intervention.
Time Frame: At baseline and post-intervention (~4-5 weeks after first visit)
Population: as for outcome 3
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Concentration of Heat Shock Protein 25
Description: Serum levels of heat shock proteins (HSP25) will be measured via Western blots and Elisa assays in serum at baseline and post-intervention.
Time Frame: At baseline and post-intervention (~4-5 weeks after first visit)
Population: as for outcome 3
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Concentration of Heat Shock Protein Transcription Factor 1
Description: Serum levels of heat shock protein transcription factor (HSF1) will be measured via Western blots and Elisa assays in serum at baseline and post-intervention.
Time Frame: At baseline and post-intervention (~4-5 weeks after first visit)
Population: as for outcome 3
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 0

8. Secondary Outcome: Utah Early Neuropathy Scale (UENS)
Description: The Utah Early Neuropathy Scale (UENS) is a physical examination scale specific to early sensory predominant polyneuropathy. The UENS emphasizes severity and spatial distribution of pin (sharp) sensation loss in the foot and leg and focuses less on motor weakness. The UENS includes five subscales: motor examination (4), pin sensation (24), allodynia/hyperesthesia (2), large fiber sensation(8) and deep tendon reflexes (4). The UENS total score ranges from 0-42, with a low score indicating a normal neurological exam and a higher score indicating neuropathy.
Time Frame: At baseline and post-intervention (~4-5 weeks after first visit)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Heat Therapy Treatment
Number analyzed (Participants) | 2
score on a scale | 2 [1 to 3]

ADVERSE EVENTS:
Time Frame: Adverse event data would have been collected between date of enrollment through study completion, approximately 11 to 13 weeks.
Arm/Group | Heat Therapy Treatment
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
We were able to enroll 3 subjects, though 1 was a screen fail and unable to start intervention. Unfortunately recruitment was difficult due to 1) troubles identifying the population target (pre-diabetic with idiopathic neuropathy), 2) strict timing requirements of the study and 3) potential subject concerns regarding the COVID pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT05070741/Prot_SAP_000.pdf